CLINICAL TRIAL: NCT01365897
Title: Effectiveness of Modafinil in Improving Mnesic Performance and Executive Functions of University Students From Careers of High Academic Performance
Brief Title: Effectiveness of Modafinil in Improving Cognitive Performance of University Students
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Alejandro Fernández, Universidad de Valparaiso
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 04/2010
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2010-11

CONDITIONS: Attention; Memory, Short-Term; Executive Function
Keywords: Modafinil; Memory; Executive Functions; Memory, Short-Term; Attention; University Students; Stroop Effect; Digit Span; Backwards Digit Span; Biber Cognitive Estimation Test
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Control Group
  Interventions: Drug: Modafinil
- Modafinil 200mg (Experimental): Modafinil 200mg taken orally.
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — Modafinil 200mg
  Other Names: Modafinilo

SUMMARY:
The purpose of this study is to determine whether modafinil is effective in the improvement of mnesic performance and executive functions of university students from high academic performance.

ELIGIBILITY:
Inclusion Criteria:

* Medicine, Psychology, Obstetrics, Nursing and Kinesiology students of the Universidad de Valparaiso.

Exclusion Criteria:

* Patients with Mental Disorders.
* Patients with physical diseases.
* Patients using any psychotropic substances.
* History of chronic diseases.
* Pregnant women.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Average Correct Answers in Biber Cognitive Estimation Test | 2 hours after pill ingestion
Average response latency in Stroop Effect test | 2 hours after pill ingestion
Average Score in Digit Span test | 2 hours after pill ingestion
Average Score in Backwards Digit Span test | 2 hours after pill ingestion
Average percentage of correct answers in Stroop Effect test | 2 hours after pill ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Fernández, Psychologist, Principal Investigator — Universidad de Valparaiso; Eva Madrid, PhD, Study Director — Universidad de Valparaiso; Andrés Painel, BM BCh, Study Director — Universidad de Valparaiso; Jonathan Norambuena, BM BCh, Study Director — Universidad de Valparaiso; Franco Mascayano, Psychologist, Study Director — Universidad de Valparaiso; Walter Lips, Psychiatrist, Study Director — Universidad de Valparaiso; Ortega Alonso, Psychologist, Study Director — Universidad de Valparaiso
Locations (2):
- Chile (2):
  - Escuela de Medicina, Universidad de Valparaiso, Valparaíso, Región de Valparaíso
  - Escuela de Psicología, Universidad de Valparaiso, Valparaíso, Región de Valparaíso